CLINICAL TRIAL: NCT02272634
Title: A Randomized, Double-Blind, Placebo Controlled, Multicenter 2a Study to Assess Safety, Daily Respiratory Symptoms, PK, and Biomarker Variations After Administration of Either YPL-001, or Placebo in Patients With Moderate-to-Severe COPD.
Brief Title: A Phase 2a Study to Assess Safety, Daily Symptoms, PK, and Biomarkers of YPL-001 in COPD Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yungjin Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YPL-001_YJP-130403
Record Dates: First submitted 2014-10-12; First posted 2014-10-23 (Estimated); Results first posted 2021-06-25 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2021-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Treatment A (Experimental): Multiple oral YPL-001 80 mg doses (1 x 80 mg tablet + 1 x 1 YPL-001 80 mg matching placebo tablet) are administered approximately every 12 hours under fasting conditions for 55 consecutive days.
  Interventions: Drug: YPL-001 80 mg
- Treatment B (Experimental): Multiple oral YPL-001 160 mg doses (2 x 80 mg tablets) are administered approximately every 12 hours under fasting conditions for 55 consecutive days.
  Interventions: Drug: YPL-001 160 mg
- Treatment C (Placebo Comparator): Multiple oral matching placebo (2 x 1 YPL-001 80 mg matching placebo tablets) will be administered approximately every 12 hours under fasting conditions for 55 consecutive days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: YPL-001 80 mg — twice daily [BID]
  Other Names: Treatment A
  Arms: Treatment A
Drug: YPL-001 160 mg — twice daily [BID]
  Other Names: Treatment B
  Arms: Treatment B
Drug: Placebo — twice daily [BID]
  Arms: Treatment C

SUMMARY:
This is a Phase 2a, proof-of-concept, multicenter, randomized, double-blind, double dummy, 3-treatment, parallel study, with low and high YPL 001 doses (low dose and high dose twice daily [BID]) and a placebo control in moderate to severe Chronic Obstructive Pulmonary Disease (COPD) patients.

DETAILED DESCRIPTION:
Treatments are described as follows:

Treatment A: Multiple oral YPL-001 80 mg doses (1 x 80 mg tablet + 1 x 1 YPL-001 80 mg matching placebo tablet) will be administered approximately every 12 hours under fasting conditions for 55 consecutive days. Only the morning dose will be administered on Day 56.

Treatment B: Multiple oral YPL-001 160 mg doses (2 x 80 mg tablets) will be administered approximately every 12 hours under fasting conditions for 55 consecutive days. Only the morning dose will be administered on Day 56.

Treatment C: Multiple oral matching placebo (2 x 1 YPL-001 80 mg matching placebo tablets) will be administered approximately every 12 hours under fasting conditions for 55 consecutive days. Only the morning dose will be administered on Day 56. In all treatments, one tiotropium (Spiriva® HandiHaler®) 18 μg capsule will also be administered QD every morning prior to study drugs administration. Albuterol will be administered on an as needed basis. Each dose of Treatments A, B and C will be administered orally with approximately 240 mL of water.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and/or females, 30 to 85 years of age (inclusive).
* History of COPD for at least 12 months prior to screening.
* Diagnosed with COPD as defined by the American Thoracic Society (ATS)/European Respiratory Society (ERS) guidelines with symptoms compatible with COPD for at least 12 months prior to screening.
* Classified as moderate to severe COPD based on the current severity classification GOLD Stage 2-3 disease in terms of post-bronchodilator spirometry at screening
* etc.

Exclusion Criteria:

* History of life-threatening COPD including respiratory arrest, intensive care unit admission and/or requiring intubation.
* History of more than 2 hospitalizations for COPD within 12 months prior to screening.
* Presentation of an acute exacerbation of COPD that will be associated with increase sputum volume or change in sputum color within 4 weeks before Day 1 of the Run-in Period.
* Evidence of pulmonary heart disease, or clinically significant pulmonary hypertension.
* etc.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-06-04 (Actual); Primary Completion 2017-11-08 (Actual); Study Completion 2017-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard J Criner, MD, Principal Investigator — Temple University; Mark T Dransfield, MD, Principal Investigator — The Kirklin Clinic of UAB Hospital
Locations (4):
- United States (4):
  - UAB Lung Health Center, Birmingham, Alabama
  - Florida Pulmonary Research Institute, LLC, Winter Park, Florida
  - Aventiv Research Inc., Columbus, Ohio
  - Temple Lung Center, Temple University Hospital, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Lee KH, Woo J, Kim J, Lee CH, Yoo CG. YPL-001 Shows Various Beneficial Effects against Cigarette Smoke Extract-Induced Emphysema Formation: Anti-Inflammatory, Anti-Oxidative, and Anti-Apoptotic Effects. Antioxidants (Basel). 2022 Dec 22;12(1):15. doi: 10.3390/antiox12010015. PMID 36670877
- [Derived] Lee SU, Lee S, Ro H, Choi JH, Ryu HW, Kim MO, Yuk HJ, Lee J, Hong ST, Oh SR. Piscroside C inhibits TNF-alpha/NF-kappaB pathway by the suppression of PKCdelta activity for TNF-RSC formation in human airway epithelial cells. Phytomedicine. 2018 Feb 1;40:148-157. doi: 10.1016/j.phymed.2018.01.012. Epub 2018 Jan 31. PMID 29496167
- [Derived] Ryu HW, Lee SU, Lee S, Song HH, Son TH, Kim YU, Yuk HJ, Ro H, Lee CK, Hong ST, Oh SR. 3-Methoxy-catalposide inhibits inflammatory effects in lipopolysaccharide-stimulated RAW264.7 macrophages. Cytokine. 2017 Mar;91:57-64. doi: 10.1016/j.cyto.2016.12.006. Epub 2016 Dec 21. PMID 28011397
- [Derived] Lee SU, Sung MH, Ryu HW, Lee J, Kim HS, In HJ, Ahn KS, Lee HJ, Lee HK, Shin DH, Lee Y, Hong ST, Oh SR. Verproside inhibits TNF-alpha-induced MUC5AC expression through suppression of the TNF-alpha/NF-kappaB pathway in human airway epithelial cells. Cytokine. 2016 Jan;77:168-75. doi: 10.1016/j.cyto.2015.08.262. Epub 2015 Aug 28. PMID 26318254

RESULTS

PARTICIPANT FLOW:
Groups:
- YPL-001 Low Dose: Active arm including patients who receive the YPL-001 low dose. YPL-001 low dose: twice daily [BID]
- YPL-001 High Dose: Active arm including patients who receive the YPL-001 high dose, YPL-001 high dose: twice daily [BID]
- Placebo: Control arm including patients who receive the placebo drug. Placebo: twice daily [BID]
Period: Overall Study
Arm/Group | YPL-001 Low Dose | YPL-001 High Dose | Placebo
Started | 20 | 21 | 20
Completed | 19 | 20 | 19
Not Completed | 1 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All available data for patients who received at least one dose of the investigational product (i.e., YPL-001) or placebo.
Groups:
- Treatment A: Multiple oral doses of YPL-001 80 mg BID on Days 1 - 55 and QD on Day 56 AM
- Treatment B: Multiple oral doses of YPL-001 160 mg BID on Days 1 - 55 and QD on Day 56 AM
- Treatment C: Multiple oral doses of placebo BID on Days 1 - 55 and QD on Day 56 AM
- Total: Total of all reporting groups
Arm/Group | Treatment A | Treatment B | Treatment C | Total
Number analyzed (Participants) | 20 | 21 | 20 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (8.66) | 60.4 (6.50) | 61.7 (7.95) | 62.6 (7.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 9 | 25
  Male | 12 | 13 | 11 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 19 | 21 | 20 | 60
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 6 | 5 | 16
  White | 15 | 15 | 15 | 45
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 21 | 20 | 61
Body mass index [Mean (Standard Deviation); unit: kg/m²] | 28.34 (4.759) | 27.77 (3.838) | 26.19 (4.711) | 27.44 (4.465)

OUTCOME MEASURES:

1. Primary Outcome: Treatment-Emergent Adverse Event Frequency by Treatment - Number of Patients Reporting Events
Description: A TEAE was defined as an AE that was starting or worsening at the time of or after study drug administration. All AEs collected by the clinics and recorded in the CRF were captured in the database and were listed in by-patient data listings.
Time Frame: Up to Day 56
Population: All available data for patients who received at least one dose of the investigational product (i.e., YPL-001) or placebo. Safety data for all discontinued patients included in this set for the time points for which their data are available.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 20 | 21 | 20
Participants
  Number of Patients With AEs | 10 | 8 | 14
  Number of Patients Without AEs | 10 | 13 | 6

2. Primary Outcome: Treatment-Emergent Adverse Event Frequency by Treatment - Adverse Events
Description: as for outcome 1
Time Frame: Up to Day 56
Population: as for outcome 1
Measure: Number; unit: Adverse events
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 20 | 21 | 20
Adverse events
  Total Number of AEs | 18 | 14 | 23
  Eye disorders | 1 | 1 | 0
  Gastrointestinal disorders | 3 | 1 | 1
  Infections and infestations | 5 | 3 | 6
  Injury, poisoning and procedural complications | 0 | 0 | 2
  Metabolism and nutrition disorders | 1 | 0 | 0
  Musculoskeletal and connective tissue disorders | 1 | 2 | 0
  Nervous system disorders | 0 | 1 | 0
  Respiratory, thoracic and mediastinal disorders | 5 | 4 | 13
  Skin and subcutaneous tissue disorders | 0 | 1 | 1
  Surgical and medical procedures | 1 | 1 | 0
  Vascular disorders | 1 | 0 | 0

3. Primary Outcome: Treatment-Emergent Adverse Event Frequency by Treatment, Severity, and Relationship to Drug - Number of Patients Reporting Events
Description: When a patient experienced the same AE at more than one level of severity, the patient was counted once under the highest severity.
Time Frame: Up to Day 56
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 20 | 21 | 20
participants
  Number of Patients With AEs | 10 | 8 | 14
  Severity: Mild | 3 | 3 | 4
  Severity: Moderate | 7 | 5 | 9
  Severity: Severe | 0 | 0 | 1
  Relationship to Drug: Unrelated | 9 | 7 | 14
  Relationship to Drug: Unlikely | 0 | 1 | 0
  Relationship to Drug: Possible | 1 | 0 | 0
  Relationship to Drug: Probable | 0 | 0 | 0
  Relationship to Drug: Definite | 0 | 0 | 0

4. Primary Outcome: Treatment-Emergent Adverse Event Frequency by Treatment, Severity, and Relationship to Drug - Adverse Events
Description: as for outcome 3
Time Frame: Up to Day 56
Population: as for outcome 1
Measure: Number; unit: Adverse events
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 20 | 21 | 20
Adverse events
  Number of Adverse Events | 18 | 14 | 23
  Severity: Mild | 9 | 8 | 11
  Severity: Moderate | 9 | 6 | 11
  Severity: Severe | 0 | 0 | 1
  Relationship to Drug: Unrelated | 17 | 12 | 23
  Relationship to Drug: Unlikely | 0 | 2 | 0
  Relationship to Drug: Possible | 1 | 0 | 0
  Relationship to Drug: Probable | 0 | 0 | 0
  Relationship to Drug: Definite | 0 | 0 | 0

5. Secondary Outcome: Change From Baseline in Main Peak Expiratory Flow (PEF) Measured Daily
Description: The PEF assessments are made daily prior to each dose from Day 1 of the Run-in Period to Day 56 of the Treatment Period. Three measurements were made at each time point using a hand held PEF meter. Readings not performed in the clinical research unit (CRU) were recorded in the patient e-diary. All PEF assessments were performed before administration of a bronchodilator where possible. Baseline is Day 1 predose measurement.
Time Frame: Baseline to Day 55
Population: Analysis population included data obtained from all the subjects who were enrolled in the study and received at least one dose of the investigational drug and had primary efficacy endpoint after administration of the investigational drug
Measure: Mean (Standard Deviation); unit: L/min
Groups:
- Treatment A: Multiple oral doses of YPL-001 80 mg BID on Days 1 - 55
- Treatment B: Multiple oral doses of YPL-001 160 mg BID on Days 1 - 55
- Treatment C: Multiple oral doses of placebo BID on Days 1 - 55
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 19 | 21 | 20
L/min
  Baseline (Day1): number analyzed (Participants) | 17 | 21 | 19
  Baseline (Day1) | 250.0 (109.82) | 254.9 (68.61) | 240.7 (68.21)
  Day55: number analyzed (Participants) | 17 | 17 | 16
  Day55 | 282.8 (123.61) | 277.9 (92.08) | 247.6 (96.17)

6. Secondary Outcome: Change From Baseline of Symptom Severity Score for Symptoms of Chronic Obstructive Pulmonary Disease (COPD) Exacerbation
Description: Patient is asked to record the major (sputum quality, color, consistency) and minor (cough, wheeze, sore throat, nasal congestion, discharge, and body temperature above 100°F) symptoms of COPD exacerbation via the e-diary before each dosing. Baseline is Day 1 predose measurement
  1. Breathlessness(Dyspnea) Screen: 0(None)-10(Extreme): 0: better condition, 10: worse condition
  2. Sputum Quantity Screen: None(better)-greater than 1/4 cup(worse)
  3. Sputum Color Screen: White(better)-Brown(condition)
  4. Sputum Consistency Screen: Watery(better)-Thick(worse)
  5. Peak Flow Measurement Screen: 60(better)-800(worse)
  6. Symptoms Screen: (Temperature over 100F / Cough/Wheeze/Sore Throat/ Nasal Congestion)
  7. Nasal Discharge Screen(Yes/No) * quantitative data were summarized including sample size, arithmetic mean, standard deviation, CV, min and max.
  Symptom score catecorizes normal(0-0.5), mild(1-1.5), moderate(2-2.5), severe(3-3.5)
Time Frame: Baseline to Day 55
Population: All available data for patients who received at least one dose of the investigational product (i.e., YPL-001) or placebo. Symptom monitoring data for all discontinued patients were included in this set for the time points for which their data are available.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 19 | 21 | 20
score on a scale
  Baseline (Day 1): number analyzed (Participants) | 15 | 18 | 18
  Baseline (Day 1) | 0.63 (0.812) | 0.17 (0.297) | 0.47 (0.757)
  Day 55: number analyzed (Participants) | 17 | 17 | 16
  Day 55 | 0.26 (0.504) | 0.18 (0.351) | 0.50 (0.876)

7. Secondary Outcome: Change From Baseline in Dyspnea (Modified Borg Dyspnea Scale)
Description: Severity level of patient's dyspnea is accessed via the modified Borg dyspnea scale programmed within the e-diary. The modified Borg dyspnea scale is a self-administered categorical scale with a score from 0 to 10, where 0 (as a measure of dyspnea) corresponds to the sensation of normal breathing (absence of dyspnea) and 10 corresponds to the patient's maximum possible sensation of dyspnea.
Time Frame: Baseline to Day 55
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 19 | 21 | 20
units on a scale
  Baseline (Day 1): number analyzed (Participants) | 17 | 21 | 19
  Baseline (Day 1) | 3.88 (1.996) | 4.05 (1.746) | 3.18 (2.512)
  Day 55: number analyzed (Participants) | 17 | 17 | 16
  Day 55 | 3.76 (2.463) | 3.88 (2.147) | 3.31 (2.323)

8. Secondary Outcome: Change From Baseline of Calculated Score From Duke Activity Status Index (DASI)
Description: Patient's functional capacity and activity status were accessed via the DASI programmed within the e-diary. DASI is a self-administered 12-item questionnaire that assesses daily activities such as personal care, ambulation, household tasks, sexual function and recreation with respective metabolic costs. Each item has a specific weight based on the metabolic cost. The final score ranges between 0 and 58.2 points.
  The higher score shows the better the functional capacity.
Time Frame: Baseline to Day 55
Population: All available data for patients who received at least one dose of the investigational product (i.e., YPL-001) or placebo. Symptom monitoring data for all discontinued patients included in this set for the time points for which their data are available.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 19 | 21 | 20
score on a scale | -0.267 (3.7696) | -2.844 (9.8016) | 1.137 (4.8336)

9. Other Pre Specified Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1)
Description: Forced expiratory volume in 1 second (FEV1) is the amount of air that can be exhaled in one second. FEV1 is measured by spirometry performed at approximately the same time of day on each visit to avoid diurnal variation. A positive change from baseline in FEV1 indicates improvement in lung function.
Time Frame: Baseline (Screen) to Day 55
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 19 | 21 | 20
L | -0.088 (0.2721) | -0.002 (0.1974) | 0.011 (0.1533)

10. Other Pre Specified Outcome: Change From Baseline in Inspiratory Capacity (IC)
Description: Inspiratory capacity (IC) is the maximum volume of air that can be inhaled into the lungs from the normal resting position after breathing out normally. IC is measured by spirometry performed at approximately the same time of day on each visit to avoid diurnal variation.
Time Frame: Baseline (Screening) to Day 55
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 19 | 21 | 20
L | -0.158 (0.3148) | -0.097 (0.4357) | -0.304 (0.4709)

11. Other Pre Specified Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second/Forced Vital Capacity (FEV1/FVC) Ratio
Description: The ratio is calculated as the amount of air expelled from the lungs in one second after a full inspiration (FEV1) divided by the volume of air that can forcibly be blown out after a full inspiration (FVC).
Time Frame: Baseline to Day 55
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 19 | 21 | 20
ratio | -1.8 (6.21) | -0.2 (4.63) | 2.0 (4.98)

12. Other Pre Specified Outcome: Transition Dyspnea Index (TDI) Focal Score
Description: Dyspnea at baseline (Day -1) will be assessed with the Baseline Dyspnea Index (BDI). This instrument has 3 domains (functional impairment, magnitude of task and magnitude of effort) with the values added for a combined focal score. Functional impairment determines the impact of breathlessness on the ability to carry out activities; magnitude of task determines the type of task that causes breathlessness, magnitude of effort establishes the level of effort that results in breathlessness. The BDI scores range from 0 (very severe impairment) to 4 (no impairment) for each domain with the baseline focal score consisting of the sum of each domain (0 to 12). Dyspnea throughout the study will be performed at the time points. The change from baseline is measured by the Transition Dyspnea Index (TDI) score which ranges from -3 (major deterioration) to +3 (major improvement) for each domain with the TDI focal score consisting in the sum of each domain (-9 to +9).
Time Frame: Baseline to Day 55
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 19 | 21 | 20
units on a scale | 2.2 (2.68) | 1.1 (2.75) | 2.9 (2.84)

13. Other Pre Specified Outcome: Change From Baseline in Chronic Obstructive Pulmonary Disease Assessment Test (CAT)
Description: The chronic obstructive pulmonary disease assessment test (CAT) is a short and simple questionnaire of 8 items completed by patients to be performed at the time points. Scores for each of the 8 items are summed to give a single, final score ranging from 0 (no impact on daily activities) to 40 (very high impact on daily activity).
Time Frame: Baseline to Day 55
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 19 | 21 | 20
units on a scale | -1.2 (6.14) | -1.3 (5.11) | 0.0 (7.38)

14. Other Pre Specified Outcome: Change in Percentage of Total Cells in Bronchoalveolar Lavage (BAL)
Description: The bronchoalveolar lavage (BAL) samples were collected at baseline and again at the completion of the study for pharmacodynamics (PD) assessments of biomarkers. BAL samples are at analyzed for total cell count (cells/mL) of white blood cell, macrophages, lymphocytes, neutrophils, and eosinophils as a percentage of total cells.
Time Frame: Baseline (Day -1) and Day 55
Population: All patients who received at least one dose of YPL-001 or placebo and provide at least one post-baseline PD measurement.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 19 | 20 | 20
percent change from baseline
  WBC: number analyzed (Participants) | 18 | 19 | 18
  WBC | 5.2 (23.16) | -2.3 (22.87) | -5.6 (21.16)
  Eosinohils: number analyzed (Participants) | 11 | 16 | 15
  Eosinohils | -50.8 (49.25) | 38.3 (150.97) | 61.2 (261.73)
  Lymphocytes: number analyzed (Participants) | 15 | 20 | 17
  Lymphocytes | 37.8 (111.26) | 2.7 (75.89) | 19.4 (121.45)
  Macrophages: number analyzed (Participants) | 15 | 18 | 18
  Macrophages | 45.9 (136.88) | 9.3 (55.48) | 59.8 (124.05)
  Neutrophils: number analyzed (Participants) | 15 | 20 | 18
  Neutrophils | 57.0 (152.70) | 83.5 (252.98) | 1.1 (106.19)

15. Other Pre Specified Outcome: Change in Concentrations of Inflammatory Marker in Bronchoalveolar Lavage (BAL)
Description: The bronchoalveolar lavage (BAL) samples are collected at baseline and again at the completion of the study for pharmacodynamics (PD) assessments of biomarkers. BAL samples are analyzed for concentrations of tumor necrosis factor (TNF)-alpha, interleukin (IL)-1β, IL-4, IL-5, IL-6, IL-8, IL-13, Myeloperoxidase (MPO), neutrophil elastase (ELA2), monocyte chemotactic protein-1 (MCP-1), myeloperoxidase(MPO), and matrix metalloproteinase-9 (MMP-9).
Time Frame: Baseline (Day -1) and Day 55
Population: All patients who received at least one dose of YPL-001 or placebo and provide at least one post-baseline PD measurement.
Measure: Mean (Standard Deviation); unit: % change from baseline
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 17 | 20 | 18
% change from baseline
  ELA2(neutrophil elastage) | 46.36 (154.476) | 714.18 (1864.367) | 155.57 (523.538)
  IL-13 | 34.47 (187.126) | 321.42 (1168.485) | 160.25 (243.317)
  IL-1ß | 79.65 (216.674) | 223.62 (618.896) | 45.43 (207.504)
  IL-4 | 11.12 (101.995) | 121.13 (258.496) | 155.36 (276.287)
  IL-5 | 49.97 (161.255) | 220.88 (523.979) | 213.86 (341.157)
  IL-6 | -7.41 (79.289) | 130.15 (354.531) | 53.48 (153.791)
  IL-8 | 50.61 (178.116) | 173.57 (600.987) | 45.40 (222.303)
  MCP-1 | 90.05 (224.213) | 155.50 (601.606) | 252.95 (816.196)
  MMP-9 | 28.38 (201.899) | 565.88 (2067.142) | 43.31 (242.912)
  MPO | 64.14 (243.237) | 275.50 (693.932) | 62.14 (199.545)
  TNF-a | 14.04 (114.456) | 268.19 (863.815) | 124.20 (266.423)

16. Other Pre Specified Outcome: Change in Percentage of Total Cells in Blood
Description: The blood samples are collected at the the time points of the study for pharmacodynamics (PD) assessments of biomarkers. The blood samples are analyzed for inflammatory markers (total and differential cell counts as absolute and percentage for neutrophils, macrophages, eosinophils and lymphocytes).
Time Frame: Baseline to Day 55
Population: All patients who received at least one dose of YPL-001 or placebo and provide at least one post-baseline PD measurement.
Measure: Mean (Standard Deviation); unit: % change from baseline
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 19 | 21 | 20
% change from baseline
  WBC: number analyzed (Participants) | 18 | 19 | 18
  WBC | 5.229 (23.1568) | -2.289 (22.8687) | -5.572 (21.1569)
  Eosinophils: number analyzed (Participants) | 17 | 19 | 18
  Eosinophils | 7.61728 (78.203389) | 20.06903 (91.240833) | 57.36857 (226.50576)
  Lymphocytes: number analyzed (Participants) | 18 | 19 | 18
  Lymphocytes | 10.21926 (35.449159) | -1.58746 (23.455210) | 14.24407 (26.363322)
  Monocytes: number analyzed (Participants) | 18 | 19 | 18
  Monocytes | 0.05858 (24.446709) | 30.65211 (65.329419) | 1.67563 (46.936967)
  Neutrophils: number analyzed (Participants) | 18 | 19 | 18
  Neutrophils | 1.62215 (24.058407) | 0.13700 (10.8890617) | -3.29570 (10.559662)

17. Other Pre Specified Outcome: Change in Concentrations of Inflammatory Marker in Plasma/Blood
Description: The blood samples are collected at the the time points of the study for pharmacodynamics (PD) assessments of biomarkers. The blood samples are analyzed for concentrations of C-reactive protein (CRP), fibrinogen, TNF-α, IL-1β, IL-4, IL-5, IL-6, IL-8, IL-13, MCP-1, and MMP-9. Baseline is Day 1 predose measurement.
Time Frame: Baseline to Day 55
Population: All patients who received at least one dose of YPL-001 or placebo and provide at least one post-baseline PD measurement.
Measure: Mean (Standard Deviation); unit: % change from baseline
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 19 | 21 | 20
% change from baseline
  ELA2: number analyzed (Participants) | 16 | 20 | 19
  ELA2 | -7.13 (30.726) | -17.01 (33.050) | -26.33 (30.972)
  IL-13: number analyzed (Participants) | 16 | 20 | 19
  IL-13 | 5.158 (45.4151) | 10.197 (53.7029) | -1.622 (5.5691)
  IL-1ß: number analyzed (Participants) | 16 | 20 | 19
  IL-1ß | 44.9813 (149.88595) | 32.7901 (121.71539) | 4.7453 (72.39394)
  IL-4: number analyzed (Participants) | 16 | 20 | 19
  IL-4 | 68.849 (280.7619) | 22.678 (98.3923) | -19.865 (35.6127)
  IL-5: number analyzed (Participants) | 16 | 20 | 19
  IL-5 | 73.36 (214.724) | 20.57 (257.416) | -5.30 (99.117)
  IL-6: number analyzed (Participants) | 16 | 20 | 19
  IL-6 | -26.0682 (36.92257) | -35.8383 (82.30541) | -48.4230 (51.59468)
  IL-8: number analyzed (Participants) | 16 | 20 | 19
  IL-8 | 26.916 (47.0832) | 6.986 (54.7421) | 57.464 (176.8141)
  MCP1: number analyzed (Participants) | 16 | 20 | 19
  MCP1 | 20.019 (86.8398) | -13.923 (31.9128) | 51.441 (173.5531)
  MMP9: number analyzed (Participants) | 16 | 20 | 19
  MMP9 | -10.922 (52.3542) | -9.087 (39.4842) | -27.524 (34.8440)
  MPO: number analyzed (Participants) | 16 | 20 | 19
  MPO | -6.051 (21.3202) | -9.661 (26.7605) | -14.232 (26.6217)
  TNF-α: number analyzed (Participants) | 16 | 20 | 19
  TNF-α | -10.499 (24.7753) | -16.184 (25.6551) | -1.585 (27.5520)
  CRP: number analyzed (Participants) | 16 | 19 | 19
  CRP | -12.087 (102.3304) | 29.028 (345.0216) | -61.732 (40.0405)
  Fibrinogen: number analyzed (Participants) | 15 | 19 | 19
  Fibrinogen | 0.5 (15.39) | -0.4 (13.88) | -7.7 (22.38)

18. Other Pre Specified Outcome: Number of Participants With COPD Exacerbation
Description: Number of COPD exacerbation during 8-week treatment. COPD exacerbations are defined as a new onset or worsening of at least one respiratory symptom (i.e. dyspnea, cough, sputum purulence or volume, or wheeze) present for at least 3 consecutive days, documented change or increase in COPD-related treatment due to worsening symptoms or documented COPD-related hospitalizations or emergency room visits.
Time Frame: Baseline to Day 56
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 20 | 21 | 20
Participants | 3 | 2 | 5

19. Other Pre Specified Outcome: Change From Baseline in Forced Vital Capacity (FVC)
Description: Forced vital capacity (FVC) is the volume of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. FVC is measured by spirometry performed at approximately the same time of day on each visit to avoid diurnal variation. A positive change from baseline in FVC indicates improvement in lung function.
Time Frame: Baseline (Screen) to Day 55
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 19 | 21 | 20
L | -0.087 (0.3475) | 0.007 (0.2290) | -0.105 (0.3117)

ADVERSE EVENTS:
Time Frame: 56 days
Arm/Group | Treatment A | Treatment B | Treatment C
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 1/20
Other Adverse Events (participants affected / at risk) | 10/20 | 8/21 | 14/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=20) | Treatment B (N=21) | Treatment C (N=20)
Acute Exacerbation of COPD (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=20) | Treatment B (N=21) | Treatment C (N=20)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Skeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Large intestinal polypectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-06-08): https://cdn.clinicaltrials.gov/large-docs/34/NCT02272634/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/34/NCT02272634/SAP_001.pdf